CLINICAL TRIAL: NCT06452953
Title: Comparative Study on the Cognitive Function and Brain Imaging of Modified Suanzaoren Decoction and Eszopiclone in the Treatment of Primary Insomnia Patients With Yin Deficiency and Hyperactivity of Fire Syndrome
Brief Title: Modified Suanzaoren Decoction Versus Eszopiclone for the Treatment of Chronic Insomnia Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: The Third Hospital of Inner Mongolia Autonomous Region (Unknown)
Responsible Party: Principal Investigator, Guo Wenbin, Professor of Psychiatry Department of Psychiatry of the Second Xiangya Hospital, Central South University, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019MS08099
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Chronic Insomnia Disorder
Keywords: suanzaoren decoction; eszopiclone; polysomnography
MeSH Terms: interventions — Eszopiclone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suanzaoren decoction (Experimental): The modified Suanzaoren decoction consists of 30.0g of jujube kernel, 15.0g of Chuanchang rhizome and poria, 3.0g of licorice, and 3.0g of amber. It is administered once in the morning and once in the evening.
  Interventions: Drug: suanzaoren decoction
- eszopiclone (Active Comparator): Eszopiclone: Take 1mg nightly before bedtime.
  Interventions: Drug: Eszopiclone 1 mg

INTERVENTIONS:
Drug: suanzaoren decoction — The Suanzaoren decoction is a Chinese herbal formula known for nourishing the blood, calming the mind, and nourishing the heart and liver
  Other Names: Suan Zao Ren Tang
  Arms: suanzaoren decoction
Drug: Eszopiclone 1 mg — Eszopiclone is used in the treatment of various types of insomnia.
  Other Names: Estorra
  Arms: eszopiclone

SUMMARY:
The purpose of this study is to observe the cognitive function and clinical efficacy of modified Suanzaoren decoction and eszopiclone in the treatment of chronic insomnia disorder patients, and to investigate the possible neural mechanisms using MRI techniques.

DETAILED DESCRIPTION:
The subjects were enrolled and divided into two treatment groups using the randomized numeric table method. Each group received either modified Suanzaoren decoction or eszopiclone treatment for a period of 4 weeks. General demographic data were collected, and changes in sleep, mood, cognitive function, and rs-fMRI before and after treatment were observed. Assessment tools included the Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI), Hamilton Anxiety Scale (HAMA), and Hamilton Depression Scale (HAMD) for subjective measures, as well as the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and polysomnography (PSG) for objective evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Have adequate comprehension ability, with at least 9 years of education.
* Western medical diagnosis criteria (meeting the diagnostic criteria for chronic insomnia disorder in ICSD-3).
* Patient's subjective dissatisfaction with either the total duration or quality of sleep: difficulty falling asleep, difficulty maintaining sleep, or early awakening.
* Frequency of sleep problems: occurring at least 3 nights per week, and persisting for at least 3 months.

Exclusion Criteria:

* Individuals who have used sedatives or hypnotics, or psychiatric medications in the week prior to enrollment.
* Individuals who regularly consume strong tea, have a high smoking volume, or are dependent on coffee.
* Women who are pregnant or breastfeeding.
* Patients with severe primary diseases such as severe cardiovascular and cerebrovascular diseases, other mental disorders, or severe obstructive sleep apnea syndrome.
* Individuals with allergies or multiple drug allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The improvement of insomnia before and after treatment was assessed using the Pittsburgh Sleep Quality Index | 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire that assesses sleep quality and disturbances over a one-month time interval. It consists of 19 items that generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.

SECONDARY OUTCOMES:
The sleep condition before and after treatment is reflected using polysomnography | 4 weeks
  Polysomnography is a comprehensive test used to diagnose sleep disorders. It records various body functions during sleep, including brain waves, eye movements, muscle activity, heart rhythm, and breathing patterns. This information helps clinicians evaluate sleep quality and diagnose sleep disorders such as sleep apnea, insomnia, and REM behavior disorder.
The depression condition before and after treatment is evaluated by Hamilton Depression Rating scale | 4 weeks
  The Hamilton Depression Rating Scale is a widely used tool to measure the severity of depression in individuals. It consists of 17 items that assess various symptoms of depression, such as mood, guilt, suicidal thoughts, and sleep disturbances. Each item is scored based on the severity of the symptom, and the total score indicates the overall severity of depression, with higher scores indicating more severe depression.
The anxiety condition before and after treatment is evaluated by Hamilton Anxiety Rating scale | 4 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) is a widely used tool for assessing the severity of anxiety symptoms in individuals. It consists of 14 items that measure various aspects of anxiety, including psychological, physical, and behavioral symptoms.
The cognition function before and after treatment is evaluated by Repeatable Battery for the Assessment of Neuropsychological Status | 4 weeks
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a widely used neuropsychological assessment tool designed to evaluate cognitive function across various domains. It consists of 12 subtests that assess attention, language, visuospatial/constructional abilities, and immediate and delayed memory.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Guo, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, China

REFERENCES:
- [Derived] Yao P, Guo X, Guo Z, Lin W, Liu M, Chen M, Li J, Cui LB, Lv D. Clinical efficacy of modified suanzaoren decoction compared to esazolam tablets in the treatment of chronic insomnia disorder. Front Psychiatry. 2025 Jul 24;16:1533652. doi: 10.3389/fpsyt.2025.1533652. eCollection 2025. PMID 40778328
- [Derived] Zhang L, Guo Z, Han Y, Yan H, Lv D, Yao P, Zhao J, Chen L, Guo W. Altered cerebral functional activity and its associated genetic profiles underlying chronic insomnia disorder before and after treatment. World J Biol Psychiatry. 2025 Jun;26(5):211-223. doi: 10.1080/15622975.2025.2503938. Epub 2025 May 18. PMID 40384005